CLINICAL TRIAL: NCT00235027
Title: Improving Safety By Computerizing Outpatient Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, david bates, Chief of General Internal Medicine, BWH, Agency for Healthcare Research and Quality (AHRQ)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RO1 HS 11169
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Impact of Electronic Prescribing on Medication Safety

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- Adverse Drug Event Monitoring (Experimental): In this intervention arm, clinicians received medication safety alerts when they prescribed medications in the electronic medical record.
  Interventions: Other: Adverse Drug Event Monitoring
- Care as Usual (No Intervention): In this arm, clinicians did not receive the medication safety alerts.

INTERVENTIONS:
Other: Adverse Drug Event Monitoring — The intervention in this study is the presentation of medication safety alerts in the electronic medical record to improve patient outcomes and safety.
  Arms: Adverse Drug Event Monitoring

SUMMARY:
Patient safety is at the forefront of critical issues in health care. Medications are the single most frequent cause of adverse events, and in the inpatient setting adverse drug events (ADEs) are common, expensive, injurious to patients, and often preventable. Relatively little, however, is known about the frequency of ADEs in the ambulatory setting, how to monitor for outpatient ADEs, or on the impact of prevention strategies such as computerization of prescribing supplemented by decision-support.

DETAILED DESCRIPTION:
Specific Aim 1: Increase routine identification of outpatient adverse drug events (ADEs) through development of a computerized ADE detection monitor.

Specific Aim 2: Use basic computerized outpatient prescribing to reduce preventable ADEs in a diverse array of outpatient settings.

Specific Aim 3: Use advanced decision-support within computerized prescribing to reduce the frequency of preventable ADEs, medication errors, and potential ADEs.

ELIGIBILITY:
Inclusion Criteria: At Brigham & Women's Hospital, clinics utilizing the electronic medical record will be included. At Regenstrief, any clinic that has access to their electronic medical record will be utilized.

* For the impact of basic decision support, clinics were not randomized
* For impact of advanced decision support, clinics were randomized to receive the intervention

Exclusion Criteria:

* Clinics not using electronic medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2000-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Preventable Adverse drug events | 8/5/2004 - 1/5/2005
  Data were electronically collected each time a physician entered a prescription that triggered an alert related to medication safety.

SECONDARY OUTCOMES:
Total adverse drug events, medication errors | 1/15/2001 - 5/15/2001

CONTACTS AND LOCATIONS:
Overall Officials: Tejal K Gandhi, MD, MPH, Study Director — Brigham and Women's Hospital; David Bates, MD, Principal Investigator — Brigham and Women's Hospital; Marc Overhage, MD, Study Director — Regenstrief Institute, Inc.
Locations (2):
- United States (2):
  - Regenstrief/Indiana University, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Shah NR, Seger AC, Seger DL, Fiskio JM, Kuperman GJ, Blumenfeld B, Recklet EG, Bates DW, Gandhi TK. Improving acceptance of computerized prescribing alerts in ambulatory care. J Am Med Inform Assoc. 2006 Jan-Feb;13(1):5-11. doi: 10.1197/jamia.M1868. Epub 2005 Oct 12. PMID 16221941
- [Result] Gandhi TK, Seger AC, Overhage JM, Murray MD, Hope C, Fiskio J, Teal E, Bates DW. Outpatient adverse drug events identified by screening electronic health records. J Patient Saf. 2010 Jun;6(2):91-6. doi: 10.1097/PTS.0b013e3181dcae06. PMID 22130350
- See also: Related Info — http://www.ahcpr.gov